CLINICAL TRIAL: NCT05882708
Title: Effect of Heart Rate Control With Ivabradine on Hemodynamic in Patients With Sepsis: a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Effect of Heart Rate Control With Ivabradine on Hemodynamic in Patients With Sepsis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-LCYJ-YYDZX-02
Record Dates: First submitted 2023-05-11; First posted 2023-05-31 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Ivabradine; Hemodynamics; Heart Rate Control
MeSH Terms: conditions — Sepsis | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard treatment group (No Intervention): Standard treatment refers to that patients received active anti-infection and treatment of primary diseases according to the 2016 International Guidelines for the Management of Sepsis and septic shock. In addition, adequate volume resuscitation and vasoactive drug support can be given to maintain MAP≥65mmHg, and life support technologies such as ventilators and CRRT were given as needed.
  The target of heart rate control not mentioned in the above guidelines, was not mandatory for this group of patients with sinus tachycardia, so pharmacologic intervention was not administered.
- Ivabradine group (Experimental): Standard treatment for sepsis plus enteral ivabradine.
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — After randomization, the starting dose of ivabradine, 5mg, is given via the gastrointestinal tract every 12 hours. Heart rate control ranged from 70 to 94 bpm. Ivabradine was maintained until 96 hours after initiation of therapy. Beyond this period, the decision to continue ivabradine is left to the discretion of the treating intensivist. During the drug intervention period, heart rate is assessed before each dose. Ivabradine is tapered or discontinued if the heart rate is lower than the target rate; If the heart rate remains ≥95 bpm after 48 hours, the dose is increased to 7.5mg. If a heart rate of 95 or more bpm recurs after discontinuation during the intervention period, treatment with ivabradine can be resumed. Furthermore, Ivabradine is also discontinued at any time in the presence of severe liver impairment, malignant arrhythmia, cardiac conduction block, allergy, the need to take drugs with potentially harmful effects of ivabradine.
  Arms: Ivabradine group

SUMMARY:
Sepsis, a life-threatening syndrome, is often accompanied by tachycardia in spite of adequate volume resuscitation to correct hypovolemia and vasopressor medication to correct hypotension. Recently, relevant studies have shown that sustained tachycardia in sepsis was also related to high mortality, and appropriate control of heart rate could improve prognosis. Ivabradine reduces heart rate directly without a negative inotropic effect through inhibition of the If ionic current，which is absent from the traditional rate control drug (beta-blockers). This is a prospective, multicenter, randomized, open label study designed to compare ivabradine with placebo on the difference of heart rate and haemodynamics in patients with sepsis.

DETAILED DESCRIPTION:
This study aims to enroll 172 patients with sepsis as defined by The Third International Consensus Definitions for Sepsis and Septic Shock criteria and sinus tachycardia (HR ≥ 95 bpm) despite a hemodynamic optimization. Patients will be randomly assigned to standard treatment group (GS) or ivabradine group (GI，standard treatment for sepsis plus enteral ivabradine). Patients in GI, with a heart rate control target of 70 to 94bpm, received ivabradine within the first 96 hours after randomization, and overall participants are followed up to 28 days. The secondary outcomes include the difference in SOFA score, incidence of serious adverse events, need for organ support, length of ICU stay, and 28-day overall mortality.

Despite recent studies are limited, this study will investigate whether HR control using ivabradine is safe, feasible, and effective, and further enhance the understanding of ivabradine in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 years or above.
2. Being treated in an intensive care unit.
3. Sepsis is diagnosed according to Sepsis-3.0 criteria, which is defined as patients requiring antimicrobial agents due to confirmed or suspected infection, acute increase in the SOFA score at least 2 points.
4. Mean arterial pressure (MAP) is maintained ≥65 mmHg with adequate volume resuscitation and vasopressor therapy. Volume resuscitation is considered adequate when Central Venous Pressure (CVP) > 8mmHg, global end-diastolic volume index (GEDI) > 680ml/m2 and resting inferior vena cava (IVC) diameter > 1.5cm.
5. Patients are in a relatively stable period of hemodynamics, as defined that the targe mean arterial pressure are maintained with the same dosage of vasopressors for at least 2 h.
6. Sinus rhythm with heart rate ≥ 95bpm maintain for at least 2 hours but less than 72 hours.

Exclusion Criteria:

1. Patients who had received ivabradine therapy or known allergy to it prior to randomization.
2. Patients with severe liver dysfunction (Child-C grade).
3. Patients with a history of pre-existing chronic renal failure (glomerular filtration rate less than 15 ml/min/1.73 m2), except patients treated with continuous renal replacement therapy (CRRT).
4. Patients with known seizure disorder.
5. Patients with any contraindication to gastrointestinal drug administration.
6. Pregnant or lactating patients.
7. patients requiring the use of potent cytochrome CYP3A4 inhibitors such as antifungals of the azole-type (specifically ketoconazole and itraconazole), macrolide antibiotics (specifically clarithromycin and erythromycin) and HIV protease inhibitors (specifically nelfinavir and ritonavir).
8. Patients with active bleeding;
9. Patients with cardiac dysfunction caused by non-septic causes such as recent (< 2months) acute myocardial infarction, chronic cardiac dysfunction (NYHA Class Ⅳ), congenital heart disease, pericardial tamponade, severe aortic regurgitation and aortic coarctation before enrollment.
10. Patients with sinoatrial block, sick sinus syndrome, atrioventricular block or heart rate dependence on pacemaker.
11. Patients with refractory shock, which may be considered if one of the following conditions still exists in spite of active volume resuscitation, high doses of vasoactive drugs (VIS score >120), and other regular therapy: 1) Worsening hypotension (MAP<65mmHg); 2) Lactate persistence>5mmol/L (two times in a row with an interval of more than 30min), and a progressive upward trend; 3) Mixed venous blood oxygen saturation (SvO2) sustained <55% (more than two consecutive times, more than 30min apart), and progressive deterioration. The above conditions lasted for more than 5 hours.
12. Use of beta blockers within 24 hours before enrollment.
13. Pheochromocytoma patients.
14. After cardiopulmonary resuscitation.
15. Patients who have been enrolled in another interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The difference of a reduction in heart rate | 96 hours
  Heart rate is a continuous variable with repeated measurements during the first 96 hours after enrollment, the area under the curve (AUC) relative to baseline are calculated for each group, and then difference in AUC are compared.
The difference in MAP | 96 hours
  MAP will be recorded every 12 hours for each patient during the first 96 hours after enrollment. The area under the curve (AUC) relative to baseline are calculated for each group, and then difference in AUC are compared. The change in this index will be used to evaluate the hemodynamic effects of ivabradine.
The difference in CI | 96 hours
  Cardiac index (CI) will be recorded every 12 hours for each patient during the first 96 hours after enrollment. The area under the curve (AUC) relative to baseline are calculated for each group, and then difference in AUC are compared. The change in this index will be used to evaluate the hemodynamic effects of ivabradine.
The difference in LVEF | 96 hours
  Left ventricular ejection fraction (LVEF)，measured by bedside ultrasound, will be recorded every 12 hours for each patient during the first 96 hours after enrollment. The area under the curve (AUC) relative to baseline are calculated for each group, and then difference in AUC are compared. The change in this index will be used to evaluate the hemodynamic effects of ivabradine.
The difference in SVI | 96 hours
  Stroke volume index (SVI), obtained through PiCCO, will be recorded every 12 hours for each patient during the first 96 hours after enrollment. The area under the curve (AUC) relative to baseline are calculated for each group, and then difference in AUC are compared. The change in this index will be used to evaluate the hemodynamic effects of ivabradine.
The difference in VIS | 96 hours
  Vasopressor requirement during the trial observation (or intervention) period ought to be recorded as vasoactive inotropic score (VIS) according to the formula. The area under the curve (AUC) relative to baseline are calculated for each group, and then difference in AUC are compared. The change in this index will be used to evaluate the hemodynamic effects of ivabradine.

SECONDARY OUTCOMES:
28-day overall mortality | 28 days
  Overall survival measured from randomization to death or day 28
difference of the Sequential Organ Failure Assessment score | 96 hours
  Difference of the Sequential Organ Failure Assessment (SOFA) score (0~24) at day 1, 2, 3, 4 between groups. Higher score means more illness. SOFA score include organ function measure, which can reflect the functional status of organs.
length of ICU stay | 28 days
  average length of ICU stay will be compared
The percentage of need for organ support | 28 days
  the percentage of receipt of CRRT, vasopressors and mechanical ventilation. It can reflect the functional status of organs, especially renal and pulmonary.
length of in-hospital stay | 28 days
  average length of in-hospital stay will be compared
Incidence of adverse events | 96 hours
  The incidence of adverse events will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Zhenhui Zhang, PhD, Study Director — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng J, Wen D, Pan Z, Chen X, Kong T, Wen Q, Zhou H, Chen W, Zhang Z. Effect of heart rate control with ivabradine on hemodynamic in patients with sepsis: study protocol for a prospective, multicenter, randomized controlled trial. Trials. 2024 Oct 23;25(1):710. doi: 10.1186/s13063-024-08560-5. PMID 39443954